CLINICAL TRIAL: NCT05385640
Title: Serum Potassium as a Predictor of Clinical Outcomes in an Older Patient Cohort With Chronic Postsurgical Pain: Retrospective Analysis of A Multi-Center Prospective Database in China
Brief Title: Serum Potassium as a Predictor of Clinical Outcomes in an Older Patient Cohort With Chronic Postsurgical Pain
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); First Affiliated Hospital of Guangxi Medical University (Other); Sun Yat-sen University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Peking University People's Hospital (Other); China-Japan Friendship Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Yanhong Liu, Deputy Chief of administration, Anesthesiology, Chinese PLA General Hospital
Other Study IDs: PLAGH-CPSP-002
Record Dates: First submitted 2022-05-15; First posted 2022-05-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Potassium, Decreased Level; Postsurgical Pain, Chronic
Keywords: elderly; Chronic Postsurgical Pain; risk factors; serum potassium
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPSP group: Patients who developed chronic pain 3 months after surgery
  Interventions: Other: NO intervention
- UN-CPSP group: Patients who did not develop chronic pain 3 months after surgery
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — NO intervention

SUMMARY:
Perioperative serum potassium in patients over 65 impacts recovery, quality of life and physical functioning. While perioperative serum potassium is an important preoperative risk factor for poor surgical outcomes in older adults, the relationship between perioperative serum potassium and postsurgical pain in this population has not been investigated. The investigators hypothesized that preoperative serum potassium would be associated with greater odds of postsurgical chronic pain.

DETAILED DESCRIPTION:
This study is a secondary interim analysis of 'Perioperative Database of Chinese Elderly Patients,' an ongoing prospective observational cohort study that began in 2020 at the muti-center in China with the primary aim of complications in older adults before and after surgery. The investigators described the demographics, comorbidities, and assessment scores as n (percentage) or mean (SD), as appropriate. Unadjusted bivariate analyses included t-test or χ2 test to compare differences between minimal pain and intrusive pain at 3 months after surgery based on demographics, preoperative status, baseline pain status and perioperative serum potassium. The investigators then created a logistic regression model with the outcome of persistent pain at 3 months after surgery and serum potassiumas the main predictor, adjusting for baseline pain, surgery type and surgery part and frailty status based on the hypothesis and association. The investigators also tested for the interaction between baseline pain and serum potassiumas.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric surgical patients ≥65 years old
* Diagnosis of Chronic postsurgical pain (CPSP) CPSP was made based on the guidelines of the International Society for Pain (CPSP: ICD-11) as follows: Chronic postsurgical pain is chronic pain developing or increasing in intensity after a surgical procedure and persisting beyond the healing process, i.e. at least 3 months after surgery. The pain is either localised to the surgical field, projected to the innervation territory of a nerve situated in this area, or referred to a dermatome (after surgery/injury to deep somatic or visceral tissues). Other causes of pain including infection, malignancy etc. need to be excluded as well as pain continuing from a pre-existing pain problem. Dependent on type of surgery, chronic postsurgical pain often may be neuropathic pain.

Exclusion Criteria:

* Patients in the central nervous system group were excluded from cardiac and neurosurgery, patients in the heart injury group were excluded from cardiac surgery.
* patients who did not agree to participate in the study were excluded in all groups.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 3088 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pain trajectories after surgery (Numerical Rating Scale) | Up to 3 months postoperation
  Pain intensity was assessed using a numerical rating scale (NRS) from 0 to 10, with zero representing no pain and 10 representing worst imaginable pain. The worst pain intensity was then categorized into two groups: no or mild pain (NRS from 0 to 3) and moderate to severe pain (NRS from 4 to 10).
The Brief Pain Inventory-short form | Up to 3 months postoperation
  It measured pain location in the body; pain intensity on an 11-point numerical rating scale (NRS; 0 represents "no pain" and 10 the "worst pain imaginable"); analgesic intake; perception of analgesic relief; and pain interference with daily life on an 11-point NRS (0 "does not interfere and 10"completely interferes") indistinct dimensions (general activity, mood, walking, work, relations with others, sleep, and enjoyment of life). Higher scores represent higher levels of pain interference.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | within 30 days prior to surgery ,Up to 3 months postoperation
  The PCS consists of 13 items, and each item is answered with a numeric value between 0 and 4; 0 corresponding to "not at all", and four corresponded to "all the time". Higher scores indicate a higher level of pain catastrophizing, the Chinese version of the PCS has demonstrated a good reliability and validity (Cronbach's alpha was 0.87 and the ICC was 0.97)
The trajectories of health related quality of life(HRQoL) | within 30 days prior to surgery , 1, 3, 7, 30, 90 days postoperation
  The trajectory of HRQoL is the vector of Utility values measured with EuroQol five-dimensional questionnaire(EQ-5D-5L)taken over 3 months(days 1, 3, 7, 30, 90；Day 0 is the day of surgery). The EQ-5D-5L measures health on five domains (mobility, self-care, usual activities, pain discomfort, and anxiety-depression), and the scores will be combined using Chinese general population weights to generate a single utility or index score. Utility values for the EQ-5D range from 1.00 to -0.391, where a score of 0 and 1 are regarded as equivalent to death and 'perfect health', respectively, and a score < 0 is considered as health state that is 'worse than death'.
The Frail Scale | within 30 days prior to surgery ,Up to 3 months postoperation
  Frailty was assessed prior to surgery using the Frail Scale assessment. The Frail Scale assessment is a validated 5-item scale comprising components from the Cardiovascular Health Frailty Index and Rockwood Scale. The five components measured include fatigue, resistance, ambulation, illness and loss of weight. For each item, choose "yes" and "no", "No" is assigned 0 points, "yes" is assigned 1 point.The total score of the five items is 0-5. (zero representing no frilty and 5 representing worst imaginable frilty.) Patients were classified as frail if they scored 3 or more on the 5-point scale and not frail if they scored below 3.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Weidong, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided